CLINICAL TRIAL: NCT05729113
Title: Pain Perception by the Chronic Renal Patient at the Time of Vascular Access Cannulation - a Randomized Trial
Brief Title: Pain Perception by the Chronic Renal Patient at the Time of Vascular Access Cannulation.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Joana Sofia Dias Pereira de Sousa (Other)
Collaborators: Instituto Politécnico de Leiria (Other)
Responsible Party: Sponsor-Investigator, Joana Sofia Dias Pereira de Sousa, PhD, Instituto Politécnico de Leiria
Organization: Instituto Politécnico de Leiria (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Pain perception
Record Dates: First submitted 2023-01-24; First posted 2023-02-15 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Renal Dialysis
Keywords: Arteriovenous Fistula; Renal Insufficiency Chronic; Quality of Life; Distraction
MeSH Terms: conditions — Arteriovenous Fistula; Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Distraction technique (Experimental)
  Interventions: Behavioral: Distraction technique
- Pain monitor (No Intervention)

INTERVENTIONS:
Behavioral: Distraction technique — Distribution of an anti-stress ball before the moment of cannulation of the vascular access and instructing to place it in hand opposite the limb of the vascular access
  Arms: Distraction technique

SUMMARY:
Pain in patients under hemodialysis affects chronic renal patients' quality of life. Distraction has been effective in controlling pain induced by the insertion of needles. Once applied adequately, distraction promotes endorphins' release, with efficacy in acute pain. This study aims to evaluate pain perception while puncturing the hemodialysis device using an anti-stress ball as a distraction strategy.

ELIGIBILITY:
Inclusion Criteria:

* adults over 18 years old
* able to read and write
* vascular access by a fistula or arteriovenous prosthesis, cannulated with a 15G needle
* vascular access at least with month old

Exclusion Criteria:

* patients under 18 years
* can't be able to read and/or write
* usage of topical anesthetics before treatment
* vascular access by a fistula or arteriovenous prosthesis, cannulated with smaller or larger 15G needles
* vascular access under one-month-old

Ages: 62 Years to 77 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-09-15 (Actual)

PRIMARY OUTCOMES:
Pain perception by hemodialysis patients | 12 weeks
  Assess the perceived pain by chronic kidney disease patients at the time of vascular access cannulation for hemodialysis, by a pain scale. On the intervention group was used a distraction technique, using an anti-stress ball, at weeks 7-12. On the control group there was only the measurement of pain by scale.

CONTACTS AND LOCATIONS:
Overall Officials: Joana P Sousa, PhD, Principal Investigator — Instituto Politécnico de Leiria
Locations (1):
- Diaverum, Figueira da Foz Municipality, Portugal

IPD SHARING:
Plan to Share IPD: No